CLINICAL TRIAL: NCT03693287
Title: Personalized Versus Standardized Parenteral Nutrition for Preterm Infants With a Birth Weight Greater Than 1250 Grams: a Multicenter Randomized Phase IV Clinical Trial
Brief Title: Personalized vs Standardized PN for Preterm Infants >1250g
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedali Riuniti Ancona (Other)
Collaborators: Azienda Ospedaliera di Padova (Other); Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Virgilio Paolo Carnielli, Principal Investigator, Ospedali Riuniti Ancona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SP-PP18; 2018-004946-41 (EudraCT Number)
Record Dates: First submitted 2018-09-26; First posted 2018-10-02 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Infant,Premature; Parenteral Nutrition; Growth
Keywords: Preterm; Infant; Parenteral Nutrition; Growth
MeSH Terms: conditions — Premature Birth; Hyperphagia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients/Parents/Legal guardian will be masked. The statistician will be also masked when analyzing the data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized-Parenteral Nutrition (P-PN) (Active Comparator): These patients will receive personalized parenteral nutrition (PN) as it is customary in the participating centers.
  Dosing range: glucose from 9 to 13 g/kg/d, AA from 2.0 to 3.0 g/kg/d, and FAT from 1.5 to 2.5 g/kg/d.
  Intravenous macronutrient intakes:
  * PN day 1: 2.0 g/kg of AA, 1.6 g/kg of FAT and 9 g/kg of glucides.
  * PN day 2: 2.5 g/kg of AA, 2.0 g/kg of FAT and 11 g/kg of glucides.
  * PN day 3 and the days after: 3.0 g/kg of AA, 2.5 g/kg of FAT and 13 g/kg of glucides.
  Intravenous vitamins will be supplied according to local clinical practice. Variations in macronutrient intakes will be tolerated within ±20%.
  Nutritional goal: to ensure at least 2.5 g/kg/d of AA and 70 kcal/kg/d of no protein energy (NPE) from PN day 2.
  Interventions: Drug: Personalized-parenteral nutrition (P-PN)
- Standardized-Parenteral Nutrition (S-PN) (Experimental): These patients will receive standardized parenteral nutrition (PN) by using a triple chamber bag (Numeta G13%E®).
  Dosing range: 80-300 ml/d. Intravenous macronutrient intakes: 65 ml/kg at PN day 1, 80 ml/kg at PN day 2 and then 100 ml/kg from PN day 3.
  Nutritional goal: to ensure at least 2.5 g/kg/d of amino acids (AA) and 70 kcal/kg/d of no protein energy (NPE) from PN day 2.
  Interventions: Drug: Standardized-parenteral nutrition (S-PN)

INTERVENTIONS:
Drug: Standardized-parenteral nutrition (S-PN) — NUMETA G13%E 300 mL is a triple-chamber (lipid emulsion, amino acids solution with electrolytes, and glucose solution), ready-to-use parenteral nutrition product available to treat preterm infants (less than 37 weeks gestational age).
  Arms: Standardized-Parenteral Nutrition (S-PN)
Drug: Personalized-parenteral nutrition (P-PN) — Intravenous glucose will be "dextrose 50%", amino acids (AA) will be "Primene®" and lipids (FAT) will be "Clinoleic®".
  Parenteral nutrition bags will be prepared by the hospital pharmacy according to the prescription of the attending neonatologist.
  Arms: Personalized-Parenteral Nutrition (P-PN)

SUMMARY:
Preterm infants (gestational age between 189 and 258 days) with a birth weight (BW) greater than 1250 grams will be randomized to personalized-parenteral nutrition (P-PN) or standardized-parenteral nutrition (S-PN). The aim of the study is to evaluate the effect of S-PN versus P-PN on growth of preterm infants with BW>1250 grams.

DETAILED DESCRIPTION:
Parenteral nutrition (PN) is a crucial part of the clinical care of preterm infants. Traditionally different components of PN are prescribed individually considering requirements of an individual infant (P-PN). Recently, standardized PN formulations (S-PN) for preterm infants have been assessed and may have advantages including a better provision of nutrients, less prescription and administration errors, decreased risk of infection, and cost savings. The recent introduction of triple-chamber bags that provides total nutrient admixture for infants may have the additional advantage of decreased risk of contamination and ease of administration.

The proposed intervention and hypothesis: The investigators propose a multi-centered Phase IV RCT to compare S-PN versus P-PN, that is the usual care for preterm infants with a birth weight >1250 grams requiring PN in the intensive care units involved in the study. The investigators hypothesize that weight gain during PN of preterm infants with a BW greater than 1250 grams who received S-PN is not statically inferior (< 2g/kg/d) to that of infants who received P-PN (Non-inferiority study).

Study design: Preterm infants (gestational age between 189 and 258 days) with a BW greater than 1250 grams will be enrolled during hospitalization after the informed consent is drawn from parents or legal guardians. All infants will undergo a physical examination and the need of PN will be judged by the caring physician according to predefined criteria. Infants requiring PN will be divided into 3 clinical groups:

* Group A or EARLY HIGH-RISK INFANTS: these infants present in rather severe conditions at birth or soon after birth which make enteral nutrition (EN) impossible or non-desirable. In this group of infants, the investigators will include patients with Perinatal asphyxia, Perinatal shock (Cardiovascular or Septic), GI malformations, Severe Intra-uterine growth retardation (IUGR) with markedly abnormal prenatal doppler, and Miscellanea. These infants will have a central venous access soon after birth.
* Group B or INSUFFICIENT EN INTAKE: these Infants are in rather stable conditions after birth, however these infants may exhibit gastrointestinal (GI) intolerance of any origin. These patients will be randomized after 72 hours of life if the mean EN volume of the first 72-hrs of life will be less than 30 ml/kg/d or if EN intake on the third day will be less than 45 ml/kg/d. In this category, the investigators will include also those infants who will have their EN intake reduced below 30 ml/kg for 3 consecutive days (usually from day 3 through day 6) because of PDA treatment. These infants will have a central venous access inserted on the 3rd or 4th day of life if not already in place.
* Group C or LATE SICKNESS: these are the infants that experience a major sickness after a variable period of good gastrointestinal tolerance. In this group, the investigators will have infants with Necrotizing Enterocolitis (NEC), Severe Sepsis with abdominal distension and poor peristalsis, Septic Shock, or other severe unexpected conditions such as volvulus etc. These infants will also have a central venous access.

Study infants within each clinical group will be divided into 2 blocks on the basis of their BW: 1250-1750 g (Block A) e >1750 g (Block B). Infants of each study group will be then randomly assigned to P-PN or S-PN (Intervention-arm). The study PN bags will be used until the study infants will not be able to tolerate 135 ml/kg/d enterally (range: 120-160 ml/kg/d according to the local practice) or until day 28 of PN (after the 28th day of PN, patients will receive PN according to the normal clinical practice).

ELIGIBILITY:
Inclusion Criteria:

* Birth weight greater than 1250 grams,
* Gestational age between 189 and 258 days,
* In need of parenteral nutrition (PN),
* Signed informed consent by at least one parent or legal guardian.

Exclusion Criteria:

* Genetic, metabolic, or endocrine disorders diagnosed before/after enrolment
* Ceftriaxone or Coumarin therapy before/after enrolment,
* Calcium therapy before enrolment,
* Cholestasis or hepatic insufficiency before enrolment,
* Renal insufficiency before enrolment,
* Hyponatremia before enrolment,
* Hypertriglyceridemia before enrolment,
* Hypersensitivity reaction to components of parenteral nutrition before/after enrolment,
* Off-label use of drug therapy before/after enrolment,
* Absent informed consent.

Ages: 189 Days to 258 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2021-07-04 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
WEIGHT CHANGE | From the start to the stop of PN (endpoint: PN day 28 if PN duration >28 days). At least 7 days of PN will be required to calculate weight gain during PN.
  Daily weight change (g/kg/d) during parenteral nutrition (PN)

SECONDARY OUTCOMES:
MUSCLE ULTRASOUND (optional) | At the start of PN, after 7, 14 and 28 days (+-1 d).
  Ultrasound measurement of mid thigh and mid arm muscle thickness (cm).
ADIPOSE TISSUE ULTRASOUND (optional) | At the start of PN, after 7, 14 and 28 days (+-1 d).
  Ultrasound measurement of mid thigh and mid arm adipose tissue thickness (cm).
BONE ULTRASOUND (optional) | At the start of PN, after 7, 14 and 28 days (+-1 d).
  Metacarpus speed of sound (m/s) and metacarpus bone transmission time (ms).
WEIGHT | Daily up to 42 weeks of post menstrual age or discharge if it comes first.
  Weight measured by a digital infant scale (grams)
TOTAL BODY LENGTH | Weekly up to 42 weeks of post menstrual age or discharge if it comes first.
  Total body length measured by a neonatal stadiometer (cm)
HEAD CIRCUMFERENCE | Weekly up to 42 weeks of post menstrual age or discharge if it comes first.
  Head circumference measured by a flexible non-stretchable tape (cm)
GLUCIDE TOLERANCE | Daily from the start to the stop of PN (endpoint: PN day 28 if PN duration >28 days).
  Blood glycemia (mg/dl).
AMINO ACID TOLERANCE | At the start of PN, at PN day 7 (+-1 d) and 14 (+-1 d), and then every 2 weeks until the stop of PN (endpoint: PN day 28 if PN duration >28 days).
  Plasma and urinary urea concentrations (mg/dl).
TRIGLYCERIDE CONCENTRATION | At PN day 3 (+-1 d) and 7(+-1 d), and then every 7 days (+-1 d) until the stop of PN (endpoint: PN day 28 if PN duration >28 days).
  Plasma triglycerides (TG; mg/dl).
FATTY ACID CONCENTRATION (optional) | At PN day 7 (+-1 d).
  Plasma fatty acid concentration (FA; mg/dl).
DICARBOXYLIC AND HYDROXYL FATTY ACID CONCENTRATION (optional) | At PN day 7 (+-1 d).
  Urinary dicarboxylic acids (DCA; mmol/mol creatinine) and hydroxyl fatty acids (H-FA; mmol/mol creatinine).
ELECTROLYTE CONCENTRATION | Daily from the start to the stop of PN (endpoint: PN day 28 if PN duration >28 days).
  Hemogasanalysis (Na+, mmol/l; K+, mmol/l; Ca2+, mg/dl; Cl-, mmol/l) and SBE (standard base excess, mmol/L)
HYPER AND HYPO-NATREMIA, -KALEMIA, -CHLOREMIA, -PHOSPHATEMIA, -CALCEMIA, AND -PARATHYROIDISM | Daily from the start to the stop of PN (endpoint: PN day 28 if PN duration >28 days).
  Episodes of Hyper/Hypo Natremia, -KaIemia, -Chloremia, -Phosphatemia, -Calcemia, and -Parathyroidism (number).
METABOLIC ACIDOSIS | Daily from the start to the stop of PN (endpoint: PN day 28 if PN duration >28 days).
  SBE < -7.5 mmol/L.
BONE MINERALIZATION-1: CALCIUM and PHOSPHORUS CONCENTRATIONS | At the start of PN and at PN day 7 (+-1 d). An additional measurement will be done at PN day 28 (+-1 d) in patients requiring long term PN.
  Plasma and urinary calcium and phosphorus concentrations (mg/dl).
LIVER FUNCTION: ALP, AST, ALT AND GGT CONCENTRATIONS | At the start of PN and at PN day 7 (+-1 d). An additional measurement will be done at PN day 28 (+-1 d) in patients requiring long term PN.
  Plasma alkaline phosphatase (ALP; UI/L), aspartate transaminase (AST; UI/L), alanine transaminase (ALT; UI/L), and gamma-glutamyl transpeptidase (GGT, UI/L).
BONE MINERALIZATION-2: PTH CONCENTRATIONS | At the start of PN and at PN day 7 (+-1 d). An additional measurement will be done at PN day 28 (+-1 d) in patients requiring long term PN.
  Plasma parathormone concentrations (PTH; pg/ml).
BONE MINERALIZATION: PYD, PICP and ICTP CONCENTRATION (optional) | At the start of PN and at PN day 28 (+-1 d) (endpoint).
  Urinary pyridinoline crosslinks of collagen (Pyd; nmol/L), serum carboxyterminal propeptide of type I procollagen (PICP; ng/mL) and serum cross-linked carboxyterminal telopeptide of type I collagen (ICTP; ng/mL)
BILIRUBIN CONCENTRATION | At PN day 7 (+-1 d). An additional measurement will be performed at PN day 14 (+-1 d) in case of PN duration >14 days.
  Plasma bilirubin (total and conjugated; mg/dl)
MORBIDITY - 1 | Up to 42 weeks of post menstrual age or discharge if it comes first.
  The incidence of the main complication of prematurity (intraventricular hemorrhage of 3° and 4° grade; Periventricular leukomalacia; Patent ductus arteriosus; Retinopathy of Prematurity; Bronchopulmonary dysplasia and Sepsis).
MORBIDITY - 2 | Daily from the start to the stop of PN (endpoint: PN day 28 if PN duration >28 days).
  The incidence of Cholestasis and Renal and Hepatic Insufficiency.
MORTALITY BEFORE 42 WEEKS POST MENSTRUAL AGE | At 42 weeks of post menstrual age or discharge if it comes first.
  Death before 42 weeks post menstrual age (number).
MORTALITY DURING PARENTERAL NUTRITION | From the start to the stop of PN (endpoint: PN day 28 if PN duration >28 days).
  Death during PN (number).
ENTERAL NUTRITION INTAKES | Daily from the start of PN to day 28 of life.
  Enteral nutrition intakes (ml/kg).
PARENTERAL NUTRITION INTAKES: AMINO ACIDS | Daily from the start to the stop of PN (endpoint: PN day 28 if PN duration >28 days).
  Intravenous amino acid intakes (g/kg).
PARENTERAL NUTRITION INTAKES: LIPIDS | Daily from the start to the stop of PN (endpoint: PN day 28 if PN duration >28 days).
  Intravenous lipid intakes (g/kg).
PARENTERAL NUTRITION INTAKES: GLUCOSE | Daily from the start to the stop of PN (endpoint: PN day 28 if PN duration >28 days).
  Intravenous glucose intakes (g/kg).
PARENTERAL NUTRITION DURATION | Daily from the start to the stop of PN (endpoint: PN day 28 if PN duration >28 days).
  PN duration (days).
MECHANICAL VENTILATION | Up to 42 weeks of post menstrual age or discharge if it comes first.
  Mechanical ventilation duration and oxygen therapy duration (days).
DRUG THERAPIES | Up to 42 weeks of post menstrual age or discharge if it comes first.
  Drug therapy duration (hours).
PHARMACOECONOMICS | Up to 42 weeks of post menstrual age or discharge if it comes first.
  Healthcare costs (euro).
METABOLIC COMPLICATIONS | Up to 42 weeks of post menstrual age or discharge if it comes first.
  Number of hypertriglyceridemic episodes (plasma triglycerides>265mg/dL), hyperglycemic and hypoglycemic episodes (blood glycaemia>175 mg/dL and <40 mg/dL, respectively) and elevated urea (blood urea>100 mg/dL).

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (2):
  - Ospedali Riuniti Ancona, Ancona
  - Azienda Ospedaliera di Padova, Padua
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ehrenkranz RA, Dusick AM, Vohr BR, Wright LL, Wrage LA, Poole WK. Growth in the neonatal intensive care unit influences neurodevelopmental and growth outcomes of extremely low birth weight infants. Pediatrics. 2006 Apr;117(4):1253-61. doi: 10.1542/peds.2005-1368. PMID 16585322
- [Background] Evering VH, Andriessen P, Duijsters CE, Brogtrop J, Derijks LJ. The Effect of Individualized Versus Standardized Parenteral Nutrition on Body Weight in Very Preterm Infants. J Clin Med Res. 2017 Apr;9(4):339-344. doi: 10.14740/jocmr2893w. Epub 2017 Feb 21. PMID 28270894
- [Background] Smolkin T, Diab G, Shohat I, Jubran H, Blazer S, Rozen GS, Makhoul IR. Standardized versus individualized parenteral nutrition in very low birth weight infants: a comparative study. Neonatology. 2010;98(2):170-8. doi: 10.1159/000282174. Epub 2010 Mar 16. PMID 20234142
- [Background] Dice JE, Burckart GJ, Woo JT, Helms RA. Standardized versus pharmacist-monitored individualized parenteral nutrition in low-birth-weight infants. Am J Hosp Pharm. 1981 Oct;38(10):1487-9. PMID 6794364
- [Background] Yeung MY, Smyth JP, Maheshwari R, Shah S. Evaluation of standardized versus individualized total parenteral nutrition regime for neonates less than 33 weeks gestation. J Paediatr Child Health. 2003 Nov;39(8):613-7. doi: 10.1046/j.1440-1754.2003.00246.x. PMID 14629529
- [Background] Mutchie KD, Smith KA, MacKay MW, Marsh C, Juluson D. Pharmacist monitoring of parenteral nutrition: clinical and cost effectiveness. Am J Hosp Pharm. 1979 Jun;36(6):785-7. PMID 111548
- [Background] Kreissl A, Repa A, Binder C, Thanhaeuser M, Jilma B, Berger A, Haiden N. Clinical Experience With Numeta in Preterm Infants: Impact on Nutrient Intake and Costs. JPEN J Parenter Enteral Nutr. 2016 May;40(4):536-42. doi: 10.1177/0148607115569733. Epub 2015 Feb 5. PMID 25655621
- [Background] Namgung R, Tsang RC, Sierra RI, Ho ML. Normal serum indices of bone collagen biosynthesis and degradation in small for gestational age infants. J Pediatr Gastroenterol Nutr. 1996 Oct;23(3):224-8. doi: 10.1097/00005176-199610000-00004. PMID 8890070
- [Background] Rossi L, Branca F, Cianfarani S. Collagen cross-links and early postnatal growth in newborns with intrauterine growth retardation. Metabolism. 2000 Nov;49(11):1467-72. doi: 10.1053/meta.2000.17670. PMID 11092513
- [Background] Jones PJ, Winthrop AL, Schoeller DA, Swyer PR, Smith J, Filler RM, Heim T. Validation of doubly labeled water for assessing energy expenditure in infants. Pediatr Res. 1987 Mar;21(3):242-6. doi: 10.1203/00006450-198703000-00007. PMID 3104873
- [Background] Schoeller DA, Ravussin E, Schutz Y, Acheson KJ, Baertschi P, Jequier E. Energy expenditure by doubly labeled water: validation in humans and proposed calculation. Am J Physiol. 1986 May;250(5 Pt 2):R823-30. doi: 10.1152/ajpregu.1986.250.5.R823. PMID 3085521
- [Background] van Marken Lichtenbelt WD, Westerterp KR, Wouters L. Deuterium dilution as a method for determining total body water: effect of test protocol and sampling time. Br J Nutr. 1994 Oct;72(4):491-7. doi: 10.1079/bjn19940053. PMID 7986782